CLINICAL TRIAL: NCT03896997
Title: Recent Modalities in Laboratory Diagnosis of Von Willebrand Disease
Brief Title: Update in VWD Laboratory Diagnosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya omar mahmoud Aballah, principle investigator, Assiut University
Other Study IDs: VWDdiagnosis
Record Dates: First submitted 2019-03-27; First posted 2019-04-01 (Actual); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: VWD - Von Willebrand's Disease
MeSH Terms: conditions — von Willebrand Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The present study will focus on the investigation of the global contribution and limitations of the multimeric analysis and mutation analysis in the VWD diagnostic process.

1. To quantify the bleeding symptoms using bleeding assessment tools (BAT) which has developed by The International Society on Thrombosis and Haemostasis (ISTH) and correlate it to the diagnosis of different subtypes of VWD in Egyptian population.
2. To assess the utility of (gain of function mutant GpIbα binding) as a recent functional assay that measures VWF activity in VWD patients.
3. Clarify how the recent laboratory diagnostic modalities are required to streamline diagnosis , classification and improve treatment of VWD patients.
4. Explore how the molecular analysis can resolve many of the drawbacks and limitations of phenotyping diagnosis (in Egyptian population which not studied before).

DETAILED DESCRIPTION:
von Willebrand disease (VWD) is the most common inherited bleeding disorder caused by defects in amount, structure or function of von Willebrand factor (VWF) (1). The prevalence estimated on population studies ranges from 0.6% to 1.3%(2).VWD is classified into type 1 with partial deficiency of VWF , type 2 with qualitative defects of VWF and type 3 with complete deficiency of VWF (3) (4). In practice, distinctions between certain VWD types are not easy, difficulties may arise because patient phenotypes may vary over time, VWF mutations can have complex effects on phenotype, certain laboratory tests are inherently imprecise, and the boundary between normal and abnormal phenotypes may not be sharply defined(3) .Moreover, accurate diagnosis is difficult due to the variability of the disease, clinical expression and the difficulties in standardizing the panel of diagnostic tests(4) (5).The first level tests are the VWF antigen (VWF:Ag), VWF platelet binding (activity) and factor VIII activity (FVIII:C), whereas the second level tests include VWF collagen binding (VWF:CB), FVIII binding capacity (VWF:FVIIIB) and ristocetin-induced platelet aggregometry (RIPA) and multimeric analysis(6). The latest official classification of VWD refers to the VWF multimeric profile as an integral part of the diagnostic process (5, 7, 8). Pérez-Rodríguez et al., and his colleauges have classified the role of multimeric analysis into three different categories : 1) Great significance ; multimeric analysis was necessary to establish a clear diagnosis; 2) Concordant ; once established clear diagnosis with other tests, the multimeric analysis agreed with such diagnosis; 3) Not informative: the multimeric analysis did not provide information for the diagnosis(8). The multimer results in 54.6% of the patients of Pérez-Rodríguez A et al., showed great significance in diagnosis. The role of genetic analysis of VWF is tricky; It is not routinely indicated but it could be mandatory in some circumstances i.e., when test result would affect the patient's treatment choice and the suitable phenotypic assays are not available as in type 2N and 2B VWD (9). Nevertheless, there are several reasons for performing molecular analysis in patients phenotypically well characterized, e.g. confirm the patient's phenotypic diagnosis(9) , help in identifying the pathological mechanism behind certain defects or can guide in the choice of treatment and in counselling regarding inheritance(5). Inheritance counselling examples are: prenatal diagnosis of type 3 or severe type 1(9) and the identification of carrier status among family members which can be easily recognized once the proband's mutation(s) have been identified (10). The mutations identified in VWD type 3 are often clearly disease-causing mutations (nonsense, frame-shift and large deletions), whereas in VWD type 1, missense mutations often identified and can only be considered candidate mutations due to the lack of firm evidence of their causal effect. The approach of investigating gene mutations causing types 1 and 3 is similar and it is sophisticated as there is no particular area where mutations are identified, in contrast to VWD type 2, that requires only the evaluation of the exons encoding the specific functional domain(s) and the large majority of mutations are located in exon 28. This strategy can be applied to all type 2 VWD (2A, 2B, 2M and 2N)(table 1)(11).

VWD type 2A(IIA) 2A(IIE) 2A*(IIC) 2A(IID) 2B 2M 2M(CB) 2N* Domain A2 D3 D1-D2 CK A1 A1 A3 D'-D3 Exon 3' portion of 28 22, 25-27 and 5' portion of 28 2-17 51-52 5' portion of 28 5' portion of 28 29-32 17-25

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for VWD diagnosis or previously diagnosed with VWD

Exclusion Criteria:

* Patients with other bleeding disorders

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients referred for VWD diagnosis or previously diagnosed with VWD, in any age and any sex, in Upper Egypt
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2022-03-02 (Estimated); Study Completion 2023-10-02 (Estimated)

PRIMARY OUTCOMES:
Measurement of von willebrand factor multimers | one year
  Von willebrand factor multimers detection by electrophoresis
Von willebrand factor antigen | One year
  Measurement of amount of von willebrand factor antigen by IU

CONTACTS AND LOCATIONS:
Overall Officials: Azza M Mostafa, lecturar, Study Director — Assiut University; Aya o Mahmoud, ass. lecturar, Principal Investigator — Assiut University